CLINICAL TRIAL: NCT06819878
Title: A Phase III, Multicenter, Double-Blind, Placebo-Controlled, Treat-Through Study to Assess the Efficacy and Safety of Induction and Maintenance Therapy With RO7790121 in Patients With Moderately to Severely Active Crohn's Disease
Brief Title: A Study to Assess the Efficacy and Safety of Induction and Maintenance Therapy With Afimkibart (RO7790121) in Participants With Moderately to Severely Active Crohn's Disease
Acronym: SIBERITE-1
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GA45331; 2024-513053-69-00 (EU CTIS Number)
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Moderately to Severely Active Crohns Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1: Afimkibart (Experimental): Participants will receive afimkibart intravenously (IV) followed by afimkibart subcutaneous (SC) injection.
  Interventions: Drug: Afimkibart
- Arm 2: Afimkibart (Experimental): Participants will receive afimkibart IV followed by afimkibart SC injection.
  Interventions: Drug: Afimkibart
- Arm 3: Placebo (Placebo Comparator): Participants will receive placebo IV followed by placebo SC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Afimkibart — Afimkibart will be administered as IV infusion. Afimkibart will be administered as SC injection.
  Other Names: PF-06480605; RVT-3101; RG6631; RO7790121
  Arms: Arm 1: Afimkibart; Arm 2: Afimkibart
Drug: Placebo — Placebo matching IV afimkibart. Placebo matching SC afimkibart.
  Arms: Arm 3: Placebo

SUMMARY:
This Phase III, multicenter, double-blind, placebo-controlled treat-through study will evaluate the efficacy and safety of induction and maintenance therapy with Afimkibart (also known as RO7790121) in participants with moderately to severely active Crohn's disease (CD).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CD
* Moderately to severely active CD
* Bodyweight >= 40 kilogram (kg)
* Demonstrated inadequate response, loss of response and/or intolerance to at least one protocol-specified conventional or advanced CD therapy
* Males and females of childbearing potential must meet protocol criteria for contraception requirements

Exclusion Criteria:

* Current diagnosis of ulcerative colitis (UC) or indeterminate colitis, ischemic colitis, infectious colitis, radiation colitis, microscopic colitis
* Participant with a history of >= 3 bowel resections (> 2 missing segments of the 5 following segments: terminal ilelium, right colon, transverse colon, sigmoid and left colon, and rectum)
* Diagnosis of short gut or short bowel syndrome
* Presence of an ileostomy, colostomy or ileoanal pouch
* Participants with symptomatic bowel strictures, fulminant colitis, or toxic megacolon
* Presence of abdominal or perianal abscess
* Presence of rectovaginal, enterovaginal, high output enterocutaneous fistula, enterovesical fistulas or perianal fistulas with >3 openings
* Current diagnosis or suspicion of primary sclerosing cholangitis
* Pregnancy or breastfeeding, or intention of becoming pregnant during the study
* Any past or current evidence of cancer of gastrointestinal tract, definite low-grade or high-grade colonic dysplasia
* History of non-gastrointestinal cancer, with the exception of adequately treated non-metastatic basal cell or squamous cell skin cancer or in situ cervical cancer
* Evidence of infection with Clostridioides difficile (C. difficile; formerly known as Clostridium difficile), cytomegalovirus (CMV), human immunodeficiency virus (HIV), Hepatitis B (HBV), Hepatitis C (HCV) during screening
* Has evidence of active tuberculosis (TB), latent TB not successfully treated (per local guidance) or inadequately treated TB
* Has received protocol-specified prohibited medicines, including known exposure to any type of anti-TL1A therapy

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Clinical Remission per Crohn's Disease Activity Index (CDAI) Score | At Week 52
  Percentage of participants achieving a CDAI score of <150. The index is a weighted sum of scores on eight components: number of liquid or soft stools (stool frequency), abdominal pain, general well-being, number of complications, use of anti-diarrheal medication, presence of an abdominal mass, hematocrit, and percentage deviation from standard body weight. CDAI generally ranges from 0 to roughly 600, with higher values indicating greater activity.
Percentage of Participants with Endoscopic Response | At Week 52
  Percentage of participants achieving a decrease in Simple Endoscopic Score for Crohn's Disease (SES-CD) of >=50% from baseline. The SES-CD is a composite of four features of endoscopic activity (presence and size of ulcers, extent of ulcerated surface, extent of affected and presence and type of narrowings or stenosis) in up to five ileocolonic segments (terminal ileum, right colon, transverse colon, sigmoid and left colon, and rectum). Each feature is scored on a scale from 0 to 3, giving segment subscores of 0 to 12 points and a total SES-CD range of 0-60, with a higher value indicating greater severity.

SECONDARY OUTCOMES:
Percentage of Participants with Clinical Remission | At Week 12
  Percentage of participants achieving a CDAI score of <150. The index is a weighted sum of scores on eight components: number of liquid or soft stools (stool frequency), abdominal pain, general well-being, number of complications, use of anti-diarrheal medication, presence of an abdominal mass, hematocrit, and percentage deviation from standard body weight. CDAI generally ranges from 0 to roughly 600, with higher values indicating greater activity.
Percentage of Participants with Endoscopic Response | At Week 12
  Percentage of participants achieving a decrease in SES-CD of >=50% from baseline. The SES-CD is a composite of four features of endoscopic activity (presence and size of ulcers, extent of ulcerated surface, extent of affected and presence and type of narrowings or stenosis) in up to five ileocolonic segments (terminal ileum, right colon, transverse colon, sigmoid and left colon, and rectum). Each feature is scored on a scale from 0 to 3, giving segment subscores of 0 to 12 points and a total SES-CD range of 0-60, with a higher value indicating greater severity.
Percentage of Participants with Symptomatic Remission | At Week 12
  Percentage of participants with the daily number of liquid or very soft stools <=2.8 and the average of daily abdominal pain scores in the past week <=1, with neither being greater than baseline.
Percentage of Participants with Endoscopic Remission | At Week 12
  Percentage of participants with an SES-CD of 0 to 4 with a decrease from baseline >=2 and no subscore >1.
Percentage of Participants with Ulcer-free Endoscopy | At Week 12
  Percentage of participants with an SES-CD ulcerated surface subscore of 0.
Average of Daily Number of Liquid or Very Soft Stools in the Past Week (SF) | Baseline through Week 12
  Daily average number of liquid or very soft stools over 7 days.
Average of Daily Abdominal Pain Scores in the Past Week (APS) | Baseline through Week 12
  The average daily rating of abdominal pain in the past 7 days. The pain is assessed on a scale of 0-3 with 0 indicating no pain and 3 indicating severe pain.
Percentage of Participants with Endoscopic Remission | At Week 52
  Percentage of participants with SES-CD=0 to 4 with decrease from baseline >=2 and no subscore >1 .
Percentage of Participants with Symptomatic Remission | At Week 52
  Percentage of participants with the daily number of liquid or very soft stools <=2.8 and the average of daily abdominal pain scores in the past week <=1, with neither being greater than baseline.
Percentage of Participants with Corticosteroid-free Clinical Remission | At Week 52
  Percentage of participants with clinical remission at Week 52 and no use of corticosteroids for CD at least 8 weeks prior to Week 52.
Maintenance of Clinical Remission | At Weeks 12 and 52
  Percentage of participants with clinical remission at both Weeks 12 and 52.
Maintenance of Endoscopic Response | At Weeks 12 and 52
  Percentage of participants with endoscopic response at both Weeks 12 and 52.
Percentage of Participants with Clinical Remission and Endoscopic Remission at Week 52 | At Week 52
  Percentage of participants achieving a CDAI score of <150 and SES-CD of 0 to 4 with a decrease from baseline >=2 and no subscore >1 at Week 52.
Percentage of Participants with Ulcer-free Endoscopy | At Week 52
  Percentage of participants with an SES-CD ulcerated surface subscore of 0.
Bowel Urgency | Baseline through Week 12 and Week 52
  Bowel urgency from baseline through week 12 and week 52. Bowel urgency is a single-item self-reported assessment of sudden or immediate need to have a bowel movement in the past 24 hours. The item response is reported on a 4-point Likert scale, from "None" to "Severe."
Fatigue | Baseline to Week 12 and Week 52
  Fatigue, as measured by the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F), from baseline to Week 12 and Week 52. FACIT-F is a 13-item self-reported assessment of fatigue. Each item response option indicates the degree to which a given statement describing the level or impact of fatigue applies in the past 7 days. Response options are graded on a 5-point Likert-type scale, from "Not at all" to "Very much."
Inflammatory Bowel Disease Questionnaire (IBDQ) Score | Baseline to Week 12 and Week 52
  Change in IBDQ score from baseline to week 12 and 52. The IBDQ is a 32-item questionnaire that measures four domains: bowel symptoms (10 questions); systemic symptoms (5 questions); emotional function (12 questions); and social function (5 questions). The total score ranges from 32-224, with a higher score indicating a better quality of life.
Percentage of Participants with Clinical Remission: Among Biomarker-Defined Subgroups of Participants | At Week 12
  Percentage of participants achieving a CDAI score of <150 at Week 12 in biomarker-defined subgroups. The index is a weighted sum of scores on eight components: number of liquid or soft stools (stool frequency), abdominal pain, general well-being, number of complications, use of anti-diarrheal medication, presence of an abdominal mass, hematocrit, and percentage deviation from standard body weight. CDAI generally ranges from 0 to roughly 600, with higher values indicating greater activity.
Percentage of Participants with Clinical Remission: Among Biomarker-Defined Subgroups of Participants | At Week 52
  Percentage of participants achieving a CDAI score of <150 at Week 52 in biomarker-defined subgroups. The index is a weighted sum of scores on eight components: number of liquid or soft stools (stool frequency), abdominal pain, general well-being, number of complications, use of anti-diarrheal medication, presence of an abdominal mass, hematocrit, and percentage deviation from standard body weight. CDAI generally ranges from 0 to roughly 600, with higher values indicating greater activity.
Percentage of Participants with Endoscopic Response: Among Biomarker-Defined Subgroups of Participants | At Week 12
  Percentage of participants achieving a decrease in SES-CD of >=50% from baseline. The SES-CD is a composite of four features of endoscopic activity (presence and size of ulcers, extent of ulcerated surface, extent of affected and presence and type of narrowings or stenosis) in up to five ileocolonic segments (terminal ileum, right colon, transverse colon, sigmoid and left colon, and rectum). Each feature is scored on a scale from 0 to 3, giving segment subscores of 0 to 12 points and a total SES-CD range of 0-60, with a higher value indicating greater severity.
Percentage of Participants with Endoscopic Response: Among Biomarker-Defined Subgroups of Participants | At Week 52
  Percentage of participants achieving a decrease in SES-CD of >=50% from baseline. The SES-CD is a composite of four features of endoscopic activity (presence and size of ulcers, extent of ulcerated surface, extent of affected and presence and type of narrowings or stenosis) in up to five ileocolonic segments (terminal ileum, right colon, transverse colon, sigmoid and left colon, and rectum). Each feature is scored on a scale from 0 to 3, giving segment subscores of 0 to 12 points and a total SES-CD range of 0-60, with a higher value indicating greater severity.
Percentage of Participants with Clinical Response | At Week 12
  Percentage of participants with a decrease >=100 in CDAI from baseline.
Percentage of Participants with Symptomatic Response | At Week 12
  Percentage of participants with a decrease >=30% in both SF and APS, with neither being greater than baseline.
Overall Change in CD Symptoms | Baseline to Weeks 2, 6, 12 and 52
  Overall change in CD symptoms, as measured by the Patient Global Impression of Change (PGIC) from baseline to Weeks 2, 6, 12 and 52. PGIC measures overall change in Crohn's disease symptoms from "Much better" to "Much worse".
Overall Severity in CD Symptoms | Baseline to Weeks 2, 6, 12 and 52
  Overall severity in CD symptoms, as measured by the Patient Global Impression of Severity (PGIS) from baseline to Weeks 2, 6, 12 and 52. PGIS measures severity of Crohn's disease symptoms from "None" to "Very severe".
Change in General Well-being | Baseline through Week 52
  The average daily rating of general well-being in the past 7 days. Well-being is assessed on a scale of 0-4 with 0 indicating generally well and 4 indicating terrible.
Incidence and Severity of Adverse Events (AEs) | Up to 70 Weeks after Baseline
  Incidence and severity of AEs, including serious AEs, AEs leading to treatment discontinuation and AEs of special interest.
Percentage of Participants with a Presence of Draining Fistulas | Baseline through Week 12 and Week 52
  Fistulas will be assessed for draining or closed status, where closed fistulas will be assessed by the investigator as no longer draining.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (330):
- United States (90):
  - Digestive Health Specialists of the Southeast (Gastroenterology Associates of Dothan) - Dothan, Dothan, Alabama
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Arizona Digestive Health, P.C (ADH), Sun City, Arizona
  - University of Arizona-CATS Research Center, Tucson, Arizona
  - Valley View Internal Medicine, Garden Grove, California
  - 310 Clinical Research, Inglewood, California
  - UCSD Medical Center, La Jolla, California
  - Gastro Care Associates, Lancaster, California
  - Om Research LLC, Lancaster, California
  - United Gastroenterologists, Los Alamitos, California
  - Acclaim Clinical Research, Inc., San Diego, California
  - Kaiser Permanente, San Francisco, California
  - UCSF/Medical Center at Mount Zion, San Francisco, California
  - Rocky Mountain Gastroenterology, Littleton, Colorado
  - Peak Gastroenterology Surgery Center, Lone Tree, Colorado
  - Access Research Institute, Brooksville, Florida
  - Gastro Florida, Clearwater, Florida
  - HealthMed Clinical Center Inc., Coral Gables, Florida
  - Hi Tech and Global Research, LLC, Coral Gables, Florida
  - The Sister Life Research, Hialeah, Florida
  - NeoClinical Research, Hialeah, Florida
  - Clinical Research of Osceola, LLC, Kissimmee, Florida
  - Florida Research Institute - Lakewood, Lakewood Rch, Florida
  - LCC Medical Research Institute, LLC, Miami, Florida
  - Ambert Medical Research, Miami, Florida
  - Orlando Regional Healthcare, Orlando, Florida
  - Nodal Medical Center Research - NMC, Tampa, Florida
  - University of South Florida School of Medicine Morsani Center for Advanced Health Care, Tampa, Florida
  - Guardian Angel Research Center, LLC, Tampa, Florida
  - Theia Clinical Research Centers, LLC, Temple Terrace, Florida
  - Florida Medical Clinic - Orlando Health, Zephyrhills, Florida
  - Digestive Healthcare of Georgia, Atlanta, Georgia
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Gastroenterology Associates of Central Georgia, Macon, Georgia
  - Grand Teton Research Group, PLLC, Idaho Falls, Idaho
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Illinois Gastroenterology Group-Glenview powered by GI Alliance, Glenview, Illinois
  - GI Alliance - Gurnee, Gurnee, Illinois
  - Indiana University Health University Hospital, Indianapolis, Indiana
  - Gastroenterology Health Partners, PLLC, New Albany, Indiana
  - Kansas Gastroenterology, LLC under Clinical Trials Network, Wichita, Kansas
  - Tri-State Gastroenterology Associates, Crestview Hills, Kentucky
  - Gastroenterology Health Partners, PLLC, Louisville, Kentucky
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston University, Boston, Massachusetts
  - Michigan Center of Medical Research, Farmington Hills, Michigan
  - Gastroenterology Associates and Endoscopy Center of North Mississippi, Oxford, Mississippi
  - Delta Gastroenterology & Endoscopy Center, Southaven, Mississippi
  - Las Vegas Clinical Trials, LLC, North Las Vegas, Nevada
  - Mount Sinai Hospital - IBD Clinical Center, New York, New York
  - Lenox Hill Hospital, New York, New York
  - DiGiovanna Inst for Med Ed&Res, North Massapequa, New York
  - Queens Village Medical Care, Queens Village, New York
  - Mainstreet - Richmond Hill Clinic, Richmond Hill, New York
  - Gastroenterology Group Of Rochester, LLP, Rochester, New York
  - University of Rochester Medical Center, Rochester, New York
  - Atrium Health, Carolinas Healthcare System, Charlotte, North Carolina
  - Omega Research North Carolina, LLC, Fuquay-Varina, North Carolina
  - Monroe Biomedical Research, Monroe, North Carolina
  - Dayton Gastroenterology, Inc., Beavercreek, Ohio
  - Digestive Disease Consultants, Brunswick, Ohio
  - University of Cincinnati Hospital, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio Gastroenterology Group, Columbus, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Gastro Health- Liberty, Liberty Township, Ohio
  - Gastro Intestinal Research Institute of Northern Ohio, Westlake, Ohio
  - Central Sooner Research, Norman, Oklahoma
  - Frontier Clinical Re search, LLC, Uniontown, Pennsylvania
  - University Gastroenterology, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Gastroenterology Associates, Greenville, South Carolina
  - Gastro One, Germantown, Tennessee
  - Quality Medical Research, Nashville, Tennessee
  - Texas Clinical Research Institute, LLC, Arlington, Texas
  - Proactive El Paso,LLC, El Paso, Texas
  - Amel Med LLC, Georgetown, Texas
  - Cano Medical Center, Harlingen, Texas
  - TDDC dba GI Alliance Research, Mansfield, Texas
  - SMS Clinical Research, LLC, Mesquite, Texas
  - Gastroenterology Research of America, LLC, San Antonio, Texas
  - GI Alliance - Southlake, Southlake, Texas
  - Baylor Scott and White Medical Center, Temple, Texas
  - Tyler Research Institute, LLC, Tyler, Texas
  - Tidewater Gastroenterology Pllc T/A Gastro. Assoc. of Tidewater, Chesapeake, Virginia
  - Emeritas Research Group, Lansdowne Town Center, Virginia
  - Blue Ridge Medical Research - Gastroenterology Associates of Central Virginia, Lynchburg, Virginia
  - Gastroenterology Consultants and Endoscopy Center of Southwest Virginia, Roanoke, Virginia
  - Tidewater Physicians Multispecialty Group (TPMG) - Clinical Research Division - Williamsburg, Williamsburg, Virginia
  - The Vancouver Clinic, Vancouver, Washington
- Argentina (2):
  - Hospital Britanico, Ciudad Autonoma Bs As
  - Hospital Provincial del Centenario, Rosario
- Australia (9):
  - The Canberra Hospital, Garran, Australian Capital Territory
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - Mater Misericordiae Limited, South Brisbane, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Flinders Medical Center, Adelaide, South Australia
  - Lyell McEwin Hospital, Adelaide, South Australia
  - Northern Hospital, Epping, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
- Austria (4):
  - Medizinische Universität Innsbruck, Innsbruck
  - Universitätsklinikum St. Pölten, Sankt Pölten
  - Barmherzige Brüder Wien, Vienna
  - Medizinische Universität Wien, Vienna
- Belgium (10):
  - AZORG Campus Aalst-Moorselbaan, Aalst
  - Cliniques Universitaires St-Luc, Brussels
  - UZ Antwerpen, Edegem
  - AZ Maria Middelares, Ghent
  - AZ Sint Lucas (Sint Lucas), Ghent
  - Jessa Zkh (Campus Virga Jesse), Hasselt
  - CHC MontLégia, Liège
  - CHU de Liège (Sart Tilman), Liège
  - CHU HELORA - Hôpital de Mons - Site Kennedy, Mons
  - Vitaz, Sint-Niklaas
- Brazil (8):
  - CLIAGEN - Clinica de Atenção em Gastroenterologia, Especialidades e Nutrição, Salvador, Estado de Bahia
  - L2 Ip Instituto de Pesquisas Clinicas Ltda ME, Brasília, Federal District
  - Centro Digestivo de Curitiba, Curitiba, Paraná
  - Hospital de Clinicas de Porto Alegre X, Porto Alegre, Rio Grande do Sul
  - UNESP - Faculdade de Medicina da Universidade Estadual Paulista - Campus Botucatu, Botucatu, São Paulo
  - Centro de Pesquisa São Lucas, Campinas, São Paulo
  - CPQuali Pesquisa Clinica Ltda, São Paulo, São Paulo
  - BR Trials - Pesquisa Clínica, São Paulo, São Paulo
- Bulgaria (2):
  - MHAT St. Ivan Rilski, Gorna Oryahovitsa
  - MHAT Saint Karidad EAD, Plovdiv
- Canada (3):
  - South Edmonton Gastroenterology, Edmonton, Alberta
  - TDDA Specialty Research, Vaughan, Ontario
  - C.I.C. Mauricie, Trois-Rivières, Quebec
- Chile (3):
  - Hospital Guillermo Grant Benavente, Concepción
  - Medwal, Santiago
  - Clinica Universidad de Los Andes, Santiago
- China (25):
  - Peking University Third Hospital, Beijing
  - the First Hospital of Jilin University, Changchun
  - Third Xiangya Hospital Centrel South University, Changsha
  - West China Hospital of Sichuan University, Chengdu
  - Chongqing General Hospital, Chongqing
  - The First Affiliated Hospital Of Fujian Medical University, Fuzhou
  - The second Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - The sixth affiliated hospital of Sun Yat-Sen University, Guangzhou
  - Zhejiang Province Traditional Chinese Medical Hospital, Hangzhou
  - Sir Run Run Shaw Hospital Zhejiang University, Hangzhou
  - Anhui Provincial Hospital, Hefei
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - Huizhou Central People's Hospital, Huizhou
  - The 1st Affiliated Hospital of Nanchang Unversity, Nanchang
  - The First Affiliate Hospital of Guangxi Medical University, Nanning
  - The First Affiliated Hospital of Ningbo University, Ningbo
  - Shanghai East Hospital, Shanghai
  - Peking University Shenzhen Hospital, Shenzhen
  - Taizhou Hospital Of Zhejiang Province, Taizhou
  - The Central Hospital of Wuhan, Wuhan
  - Ren Min Hospital Affiliated Wu Han University, Wuhan
  - Wuxi People's Hospital, Wuxi
  - Zhongshan Hospital Xiamen University, Xiamen
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou
  - Zhuzhou Central Hospital, Zhuzhou
- Colombia (2):
  - Clinica del Country, Bogotá
  - Hospital Pablo Tobon Uribe, Medellín
- Borzan Polyclinic, Osijek, Croatia
- Czechia (4):
  - SurGal Clinic s.r.o., Brno
  - Nemocnice Ceske Budejovice a.s., České Budějovice
  - Gastroenterologie s.r.o., Hradec Králové
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
- Herlev Hospital, Herlev, Denmark
- CEMDOE (Centro Médico de Diabetes, Obesidad y Especialidades), Santo Domingo, Dominican Republic
- France (7):
  - CHU Amiens - Hopital Sud, Amiens
  - Hopital Nord, Marseille
  - CHU Nice - Hopital de l'Archet 2, Nice
  - CHU Bordeaux - Hôpital Haut-Lévêque, Pessac
  - Hopital Robert Debre, Reims
  - CHU de Rennes - Hopital de Pontchaillo, Rennes
  - CHU Saint Etienne - Hôpital Nord, Saint-Etienne
- Germany (8):
  - Charite - Campus Benjamin Franklin, Berlin
  - AGAPLESION Markus-Krankenhaus, Frankfurt
  - Klinik Johann Wolfgang von Goethe Uni, Frankfurt
  - Universitaetsklinikum Halle (Saale), Halle
  - Med. Hochschule Hannover, Hanover
  - Universitaetsklinikum Jena, Jena
  - Klinikum Mannheim GmbH Universitätsklinikum, Mannheim
  - Universitätsklinikum Ulm, Ulm
- Guatemala (2):
  - Celan S.A., Guatemala City
  - Medi-k, Guatemala City
- Hungary (7):
  - Bekes Varmegyei Kozponti Korhaz, dr Rethy Pal Tagkorhaz, Békéscsaba
  - Obudai Egeszsegugyi Centrum Kft., Budapest
  - Semmelweis Egyetem, Budapest
  - Pannonia Maganorvosi Centrum, Budapest
  - Clinexpert Gyongyos Kft, Gyöngyös
  - Clinfan Szolgaltato Kft., Szekszárd
  - Fejer Varmegyei Szent György Egyetemi Oktatokorhaz, Székesfehérvár
- India (7):
  - Shree Giriraj Multispeciality Hospital, Rajkot, Gujarat
  - Surat Institute of Digestive Sciences Hospitals, Surat, Gujarat
  - Amrita Institute of Medical Sciences, Kochi, Kerala
  - MIDAS Multispeciality Hospital, Nagpur (urban), Maharashtra
  - SR Kalla Memorial Gastro & General Hospital, Jaipur, Rajasthan
  - AIG Hospitals, Gachibowli, Telangana
  - Yashoda Hospitals, Secunderabad, Telangana
- Israel (3):
  - Soroka University Medical Centre, Beersheba, Negev
  - Rambam Health Care Campus, Haifa
  - Chaim Sheba Medical Center, Ramat Gan
- Italy (13):
  - A.O. Universitaria Ospedale Consorziale Policlinico Di Bari, Bari, Apulia
  - Azienda Ospedaliero-Universitaria "Renato Dulbecco" Catanzaro, Catanzaro, Calabria
  - Universita'degli Studi di Napoli Federico II, Napoli, Campania
  - Azienda Ospedaliera San Camillo Forlanini, Rome, Lazio
  - Ospedale Isola Tiberina Gemelli, Rome, Lazio
  - ASST Fatebenefratelli-Sacco, Polo "Ospedale Fatebenefratelli ed oftalmico", Milan, Lombardy
  - Asst Santi Paolo E Carlo, Milan, Lombardy
  - Fondazione IRCCS Policlinico San Matteo di Pavia, Pavia, Lombardy
  - ASST Rhodense - Ospedale di Rho, Rho, Lombardy
  - Istituto Clinico Humanitas, Rozzano (MI), Lombardy
  - IRCCS Ospedale Casa Sollievo della Soffenza, San Giovanni Rotondo, Lombardy
  - Ospedale Mauriziano Umberto I, Turin, Piedmont
  - Azienda Ospedaliero - Universitaria di Cagliari, Monserrato, Sardinia
- Japan (48):
  - Asahikawa Medical University Hospital, Asahikawa-shi, Hokkaido
  - Takamatsu Red Cross Hospital, Takamatsu, Kagawa-ken
  - Takagi clinic, Sendai, Miyagi
  - Gamagori City Hospital, Aichi
  - Nagoya City University Hospital, Aichi
  - National Hospital Organization Hirosaki General Medical Center, Aomori
  - Asahikawa City Hospital, Asahikawa-shi
  - Tsujinaka Hospital Kashiwanoha, Chiba
  - Fukuoka University Chikushi Hospital, Chikushino-shi
  - Ehime Prefectural Central Hospital, Ehime
  - Fukui Prefectural Hospital, Fukui
  - National Hospital Organization Kyushu Medical Center, Fukuoka
  - Kyushu University Hospital, Fukuoka
  - Fukuoka University Hospital, Fukuoka
  - Kurume University Hospital, Fukuoka
  - Kitakyushu Municipal Medical Center, Fukuoka
  - Hiroshima Prefectural Hospital, Hiroshima
  - Hiroshima University Hospital, Hiroshima
  - Sapporo Kosei General Hospital, Hokkaido
  - Sapporo Medical University Hospital, Hokkaido
  - Medical Corporation Sapporo IBD Clinic, Hokkaido
  - Hyogo Medical University Hospital, Hyōgo
  - Ishikawa Prefectural Central Hospital, Ishikawa
  - Kagawa Prefectural Central Hospital, Kagawa
  - Sameshima Hospital, Kagoshima
  - Yokohama City University Medical Center, Kanagawa
  - Gokeikai Ofuna Chuo Hospital, Kanagawa
  - Japanese Red Cross Kumamoto Hospital, Kumamoto
  - Sendai Kousei Hospital, Miyagi
  - Sendai Medical Center, Miyagi
  - Nagasaki University Hospital, Nagasaki
  - Okayama University Hospital, Okayama
  - Kinshukai Infusion Clinic, Osaka
  - National Hospital Organization Osaka National Hospital, Osaka
  - Saga-ken Medical Centre Koseikan, Saga
  - Saga University Hospital, Saga
  - National Hospital Organization Shizuoka Medical Center, Shizuoka
  - Hamamatsu University Hospital, Shizuoka
  - Matsuda Hospital, Shizuoka
  - Institute of Science Tokyo Hospital, Tokyo
  - Tokyo Metropolitan Bokutoh Hospital, Tokyo
  - Keio University Hospital, Tokyo
  - National Center for Global Health and Medicine, Tokyo
  - JCHO Tokyo Yamate Medical Center, Tokyo
  - Toyama University Hospital, Toyama
  - Japanese Red Cross Wakayama Medical Center, Wakayama
  - Yamagata University Hospital, Yamagata
  - Yamanashi Prefectural Central Hospital, Yamanashi
- Mexico (3):
  - Boca Clinical Trials Mexico S.C. (Guadalajara), Guadalajara, Jalisco
  - Hospital General de Mexico, Mexico, Tlaxcala
  - Medical Care & Research SA de CV, Mérida, Yucatán
- Netherlands (4):
  - Ziekenhuis Rijnstate, Arnhem
  - Zuyderland Medisch Centrum - Sittard Geleen, Sittard-Geleen
  - ETZ Elisabeth, Tilburg
  - Universitair Medisch Centrum Utrecht, Utrecht
- Poland (20):
  - Clinical Trials UMED Sp. z o. o., ?ód?
  - Centrum Medyczne "Medis", Bydgoszcz
  - Centrum Medyczne Lukamed Joanna Luka-Wendrowska, Chojnice
  - Endo-Med Sp. z o.o., Karczew
  - Krakowskie Centrum Medyczne - Part of Futuremeds, Krakow
  - Allmedica Badania Kliniczne Sp z o.o. Sp K., Nowy Targ
  - Wojewodzki Specjalistyczny Szpital w Olsztynie, Olsztyn
  - NZOZ Eskulap Pabianice, Pabianice
  - Trialmed CRS, Piotrkow Trybunalski
  - SOLUMED Centrum Medyczne, Późna
  - Centrum Medyczne "MEDYK", Rzeszów
  - Nowe Zdrowie-CK Kieltucki I Wspolnicy Sp. j., Staszów
  - Gastromed Sp. z o.o., Toru?
  - WIP Warsaw IBD Point Profesor Kierkus, Warsaw
  - Centralny Szpital Kliniczny MSW w Warszawie, Warsaw
  - Przychodnia EuroMediCare, Wroc?aw
  - Melita Medical, Wroc?aw
  - Vistamed & Vertigo Spó?Ka Z Ograniczon? Odpowiedzialno?Ci?, Wroc?aw
  - Centrum Medyczne Oporow, Wroclaw
  - ETG Zamosc, Zamość
- Portugal (5):
  - Hospital de Braga, Braga
  - Hospital de Santa Maria, Lisbon
  - Hospital de Sao Joao, Porto
  - Centro Hospitalar de Entre Douro e Vouga - H. São Sebastião, Santa Maria da Feira
  - Hospital Sao Teotonio, Viseu
- Puerto Rico (2):
  - Klinical Investigations Group LLC, San Juan
  - University of Puerto Rico Medical Sciences Campus, San Juan
- Serbia (6):
  - University Hospital Center Dr Dragisa Misovic - Dedinje, Belgrade
  - Clinical Hospital Center Zemun, Belgrade
  - University Hospital Medical Center Bezanijska Kosa, Belgrade
  - University Hospital Medical Center Zvezdara, Belgrade
  - Clinical Center of Vojvodina, Novi Sad
  - General Hospital "Djordje Joanovic", Zrenjanin
- Slovakia (4):
  - Cliniq s.r.o., Bratislava
  - Nemocnica Bory -Penta Hospitals, Bratislava
  - Endomed, s.r.o., Košice
  - Ustredna vojenska nemocnica SNP Ruzomberok ? FN, Ružomberok
- Spain (6):
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital de Galdakao, Galdacao, Vizcaya
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Reina Sofía, Murcia
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
  - Hospital Universitario Rio Hortega, Valladolid
- Taiwan (4):
  - National Taiwan University Hospital, Taipei, Zhongzheng District
  - E-Da Hospital, Kaohsiung City
  - Chung Shan Medical University Hospital, Taichung
  - China Medical University Hospital, Taichung
- Thailand (5):
  - Division of Gastroenterology, Depart of Medicine, Fac of Med., Chulalongkorn University, Bangkok
  - Division of Gastroenterology, Depart of Internal Med, Siriraj H, Mahidol Uni, Bangkok
  - Khon Kaen Uni, Khon Kaen
  - Thammasat University Hospital, Pathum Thani
  - Division of Gastroenterology, Depart of Medicine, Fac. of Med, Songklanagarind University, Songkhla
- United Arab Emirates (3):
  - Sheikh Shakhbout Medical City, Abu Dhabi
  - Sheikh Khalifa Medical City (SKMC), Abu Dhabi
  - Burjeel Hopital, Abu Dhabi
- United Kingdom (8):
  - Addenbrookes Hospital, Cambridge
  - St Mark's Hospital & Imperial College, Harrow
  - Royal Liverpool University Hospital, Liverpool
  - King College Hospital NHS Foundation Trust, London
  - Queen Anne Street Medical Centre, London
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - North Tyneside General Hospital, North Shields
  - Nottingham University Hospitals Queen's Medical Centre, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing